CLINICAL TRIAL: NCT07073807
Title: Mobile Health Intervention to Improve Adherence to Oral Anticancer Therapy: A Pilot Feasibility Clinical Trial
Brief Title: Mobile Health Intervention to Improve Adherence to Oral Anticancer Therapy
Acronym: SMART pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Gelareh Sadigh, Associate Professor of Radiology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 7375; UCI-25-83 (Other: University of California Irvine Chao Family Comprehensive Cancer Center)
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Neoplasms
Keywords: Cancer; Oral Anticancer Therapy; Medication Adherence; Mobile Health; Health Literacy; Symptom Management; Health-Related Social Needs; Financial Toxicity; adherence; symptom burden; reminder
MeSH Terms: conditions — Neoplasms; Medication Adherence; Financial Stress

STUDY DESIGN:
Intervention Model Description: All enrolled participants receive the SMART intervention, which includes TAPPT® smart labels for real-time OAT adherence monitoring, biweekly symptom and adherence surveys, personalized reminders, missed/extra dose management, symptom support, and monthly financial and social needs screening. There is no control or comparison arm in this single-arm feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART Intervention Arm (Experimental): Participants receive the SMART intervention, a multi-level mobile health program using TAPPT® smart labels and a web-based app for real-time OAT adherence tracking. SMART includes personalized text reminders, biweekly symptom and adherence surveys, management of missed or extra doses through oncology alerts, management of symptoms through oncology alerts or educational resources, monthly screening and support for financial and health-related social needs, and tailored educational messages for participants with low health literacy. All participants receive usual oncology care in addition to the SMART intervention.
  Interventions: Behavioral: SMART Intervention using TAPPT® for Adherence, Symptom, Financial, and Social Needs Monitoring

INTERVENTIONS:
Behavioral: SMART Intervention using TAPPT® for Adherence, Symptom, Financial, and Social Needs Monitoring — The SMART intervention uses TAPPT® smart labels and a web-based app for real-time monitoring of oral anticancer therapy adherence. It includes personalized text reminders, biweekly surveys for medication adherence and symptom burden, missed and extra dose management, symptom alerts to providers, monthly financial and health-related social needs screening with tailored resources, and educational texts for low health literacy. TAPPT® smart labels work with Android/iOS smartphones. All participants receive usual oncology care.

SUMMARY:
New oral anticancer treatments have improved survival across cancer types but introduced challenges in medication adherence and symptom management. The SMART pilot trial will test a new mobile health intervention that facilitates remote adherence and symptom monitoring, patient-provider communication outside of clinic visits regarding the use of oral anticancer treatments, and support for financial and social needs, as well as health literacy support, for 30 English- and Spanish-speaking patients. This study will increase understanding of barriers and facilitators to the use of the proposed mHealth intervention.

DETAILED DESCRIPTION:
New oral anticancer treatments (OATs) have improved survival across cancer types but introduced challenges in medication adherence and symptom management. While OATs offer convenience and at-home treatment, they involve complex dosing, drug interactions, and adverse effects requiring careful self-management, and their high out-of-pocket costs can cause financial hardship, hence resulting in suboptimal adherence. Interventions to improve OAT adherence have had mixed results. Given the widespread use of mobile technology, mobile health (mHealth) options offer scalable solutions for medication management.

It is hypothesized that an mHealth intervention offering real-time adherence tracking for any prescribed OAT, monitoring for symptoms, financial and health-related social needs (HRSNs), and providing tailored reminders, education, missed dose and symptom management, and support for financial and social needs and health literacy could improve adherence across different cancers.

This study is a 3-month single-arm trial to evaluate the feasibility and acceptability of a multi-level mHealth intervention, Supporting Medication Adherence and Resource Training (SMART), in 30 English- or Spanish-speaking patients with cancer (stratified by age < 65 and >65) with a recent prescription for OAT at Chao Family Comprehensive Cancer Center (CFCCC). All patients will use Technology-Assisted Patient-Provider Tool (TAPPT)®, a web-based app that uses smart labels with near-field communication (NFC) technology and smartphone taps to facilitate real-time adherence monitoring. This technology is adaptable to various medication package formats, compatible with both Android and iOS, and capable of monitoring multiple OATs simultaneously.

The SMART intervention includes real-time adherence monitoring, missed dose reminder and management, extra or off-cycle dose management, symptom monitoring and management, and includes financial and social needs and low health literacy support.

The study examines the feasibility and acceptability of SMART to monitor OAT adherence (Aim 1), explores the preliminary effects of SMART for patient-reported adherence, mHealth monitored adherence, patient-reported quality of life, symptom burden, and healthcare utilization at 3 months (Aim 2), and describes patients' & providers' experience with the intervention using a mixed-methods approach.

Significantly, this study will increase understanding of barriers and facilitators for using SMART intervention for a variety of OATs among English- and Spanish-speaking patients and provide preliminary data to refine our proposed intervention for a future larger randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Must speak English or Spanish
* Must be 18 years of age or older
* Have a diagnosis of any type and stage of cancer
* Have a new prescription for an oral anticancer therapy (OAT) initiated within the last 90 days or planned to start within the next 15 days
* Be receiving treatment at UCI Chao Family Comprehensive Cancer Center-affiliated oncology clinics
* Own a smartphone and be willing to receive study-related text messages.

Exclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status greater than 2
* Be medically or cognitively unable to give consent or participate in the study
* Be participating in another clinical trial that monitors adherence or symptoms related to the newly prescribed OAT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the SMART Intervention | 3 months from intervention initiation
  Feasibility will be assessed by the proportion of participants using TAPPT® adherence monitoring for the duration of therapy and the proportion completing all available biweekly surveys.
Acceptability of the SMART Intervention | 3 months from intervention initiation
  Acceptability will be measured by participant ratings on the System Usability Scale (0-100; higher scores indicating greater usability).

SECONDARY OUTCOMES:
Patient-Reported Adherence to OAT | Baseline and Biweekly through 3 months post-intervention initiation
  Patient-reported adherence assessed biweekly using the PROMIS Medication Adherence Scale (PMAS) single-item question about OAT adherence, scored on a 1-5 scale with average score transformed to 0-100. ≥80 score is considered adherent.
TAPPT®-Monitored Adherence | Continuous monitoring through 3 months post-intervention initiation
  Adherence measured by the proportion of OAT doses recorded through TAPPT® smart labels over the 3-month intervention period.
Patient-Reported Quality of Life | Baseline and 3 months post-intervention initiation
  Patient-reported QOL measured at baseline and 3 months using the PROMIS-10 Global Health instrument, scored 0-100, with higher scores indicating better QOL.
Symptom Burden | Biweekly through 3 months post-intervention initiation
  Symptom burden assessed biweekly using the MD Anderson Symptom Inventory (MDASI) severity items (0-10 scale; higher scores indicating greater symptom severity).
Financial Worry | Baseline and 3 months post-intervention initiation
  Financial worry measured using the Comprehensive Score for Financial Toxicity (COST) at baseline and 3 months; scores range from 0-44, with lower scores indicating higher financial distress.
Healthcare Utilization | 3 months from intervention initiation
  Healthcare utilization including the number of oncology office visits, urgent care/emergency department visits, and hospitalizations, collected from electronic medical records over the 3-month intervention period.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Chao Family Comprehensive Cancer Center and Ambulatory Care building, Irvine, California
  - UCI Health Cancer Center - Newport, Newport Beach, California
  - UCI Health Pacific Breast Care Center, Newport Beach, California
  - UCI Health Chao Family Comprehensive Cancer Center, Orange, California
  - UCI Health - Yorba Linda, Yorba Linda, California

IPD SHARING:
Plan to Share IPD: No